CLINICAL TRIAL: NCT00366327
Title: An Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of Bifeprunox in the Treatment of Outpatients With Schizophrenia.
Brief Title: Study Evaluating Bifeprunox in Patients With Schizophrenia.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3168A1-314; B3101010 (Other: Pfizer)
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2008-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — bifeprunox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Bifeprunox

INTERVENTIONS:
Drug: Bifeprunox — Flex dose (20 or 30 mg)tablet, QD for 1 year

SUMMARY:
An open-label extension study using a variable dose (20 to 30 mg daily) of bifeprunox to evaluate long-term safety.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients who have successfully completed Wyeth study 3168A1-313.
2. A signed and dated informed consent form for this study.
3. No major protocol violations in the previous study.

Exclusion Criteria:

1. Clinically important abnormalities in the preceding short-term study that have not resolved.
2. Use of prohibited treatments in the preceding short-term study.
3. Meeting any exclusion criteria in the preceding short-term study

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in weight from baseline/first dose of bifeprunox at each observation. | 1 year

SECONDARY OUTCOMES:
Change from baseline/first dose of bifeprunox in trigyleride levels, Positive and Negative Syndrome Scale (PANSS) score, Clinical Global Impressions (CGI) score, and waist circumference at each observation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (69):
- United States (69):
  - Little Rock, Arkansas
  - Anaheim, California
  - Boynton Beach, California
  - Buena Park, California
  - Cerritos, California
  - Costa Mesa, California
  - Escondido, California
  - Garden Grove, California
  - Glendale, California
  - Huntington Beach, California
  - La Mesa, California
  - National City, California
  - Oceanside, California
  - Paramount, California
  - Rosemead, California
  - Sacramento, California
  - San Diego, California
  - Santa Ana, California
  - Torrance, California
  - Farmington, Connecticut
  - Hartford, Connecticut
  - New London, Connecticut
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - North Miami, Florida
  - Orange City, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Coevr d'Alene, Idaho
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Joliet, Illinois
  - Naperville, Illinois
  - Indiannapolis, Indiana
  - Lake Charles, Louisiana
  - Gaithersburg, Maryland
  - Towson, Maryland
  - Pittsfield, Massachusetts
  - Worcester, Massachusetts
  - Flowood, Mississippi
  - St Louis, Missouri
  - North Platte, Nebraska
  - Cherry Hill, New Jersey
  - Clementon, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - Rochester, New York
  - Staten Island, New York
  - Butner, North Carolina
  - Morehead City, North Carolina
  - Beachwood, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - East Stroudsburg, Pennsylvania
  - Jenkintown, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Cordova, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - DeSoto, Texas
  - Houston, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Kirkland, Washington